CLINICAL TRIAL: NCT00273247
Title: Adjuvant α-Interferon Treatment After Resection of Hepatocellular Carcinoma in HCV-Related Cirrhosis: a Randomized Trial on Prevention of Cancer Recurrence
Brief Title: Treatment With IFN After Curative Resection of HCC in HCV-Related Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute, Milan (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT-98-016
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2005-09

CONDITIONS: Hepatocellular Carcinoma; Hepatitis C Virus Infection; Liver Cirrhosis; Interferon Treatment; Hepatic Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C; Liver Cirrhosis | interventions — Introns

INTERVENTIONS:
Drug: Interferon alpha-2b

SUMMARY:
We conducted a randomized controlled trial of adjuvant interferon (IFN) therapy in patients with hepatitis-C virus (HCV)-related cirrhosis who underwent curative resection of hepatocellular carcinoma (HCC) to investigate whether IFN could reduce or delay the incidence of recurrent tumor (secondary/tertiary prevention of HCC). Patients were randomly assigned to treatment with IFN (3MU thrice/wk /48 weeks) vs. no treatment after curative resection of HCC(control group)

DETAILED DESCRIPTION:
Background

Primary liver cancer (hepatocellular carcinoma, HCC) remains a major cancer-related cause of death with an estimated incidence of 1 million cases per year worldwide and particular endemic distribution related to chronic hepatitis carriers. Post-necrotic cirrhosis due to chronic infection by HBV and HCV is the leading background for HCC development with a yearly rate of 3% and a 5-year probability of survival of 20%.

Liver surgery, resection or transplantation, appears the only chance of curative treatment of the tumor, but feasibility is still ranging from 15 to 30% in Western countries at time of diagnosis. Several alternative treatments are available but their potential curative effects are lacking, due to the absence of controlled trials.

Liver resection is claimed to be feasible in order 15-30% of patients with HCC with mortality reported in major centers extremely low (5%). Technical and biological devices developed in the setting of OLT can now support the limited reserve of cirrhotic livers after resection.

Regulated segmentectomy is advisable with removal of the whole portal territory belonging to the tumor. Single nodule tumors (< 5 cm) and compensated cirrhosis (Child class A) are accepted as the best candidates for liver resection that now can be performed with minimal blood loss, and minimal ischemia damage. Intraoperative ultra sound examination is now routinely used as the golden standard for staging and detection of previously undiscovered neoplastic nodules. Hepatic decompensation with ascites development, cholestasis and variceal bleeding within three months from surgery are the main negative prognostic factors for patient survival. Five years survival exceed 50% but tumor recurrences due to cirrhosis persistence could exceed 30% after three years of follow-up. Several attempts to reduce recurrence through antiangiogenetic and antiproliferative agents have been proposed.

In the present project a prospective randomized trial of Interferon (as antiproliferative drug) versus control in anti-HCV positive patients will investigate in homogeneous categories of resected tumor possible variation in the natural history and namely a reduction of recurrence rate after curative resection.

Purpose and Study Design

The trial was intentionally designed in 1997 as an unresticted collection of patients with histologically proved HCC and a HCV-related cirrhosis selected for surgical resection of the tumor in 4 experienced surgical Liver Units in Italy. Eligible patients were stratified on the basis of concomitant anti-core antibodies against HBV (anti-HBc) into two populations: "pure HCV" (HCV-RNA:positive, anti-HBc:negative) and "mixed HCV+HBV" (HCV-RNA:positive, anti-HBc:positive). Within each strata patients were then randomized in a 1:1 ratio to treatment with α-interferon (IFN) vs. no treatment (control). No restriction criteria were applied to tumor stage, as far as the resection of HCC was judged as potentially curative at pre-operative staging, intra-operative ultrasound and post-operative pathology (clearance of surgical margins).

The study was originally designed for lymphoblastoid α-interferon; then soon after trial approval by the NCI-Milan Scientific and Ethic Committee (#98-016) the protocol was amended for allowing also the use of recombinant α-2a (Roferon-A, Hoffmann-La Roche, Nutley NJ) or α -2b interferon (Intron-A, Schering-Plough, Kenilworth, NJ). The latter was eventually the preferred form. Patients allocated to treatment received IFN 3 MU/thrice weekly for 48 weeks starting within 6 weeks from the operation. The severity of adverse events during treatment were monitored and rated. Therapy was discontinued in case of life-threatening adverse event or in case of HCC recurrence during treatment. For severe events other than anemia the IFN dose was reduced by 50%; full dose could be resumed after the event was resolved or discontinued if the effect persisted. The percentage of the total predicted dose of IFN actually assumed by each patients was recorded. Patients assuming at least 80% of the total dose of IFN and treated for at least 80% of the expected duration of therapy were a priori defined as adherent to therapy.

Recurrences were a priori defined as "early" or "late" whether or not they occurred within 2 years from the surgical removal of the HCC. In fact early recurrence were related to intra-hepatic metastases of the primary tumor possibly missed at the time of therapy, while late recurrence might be due to new cancer foci related to the persistence of HCV-related carcinogenetic factors.

Primary endpoint of this randomized clinical trial (RCT) was recurrence-free survival (RFS) while the secondary endpoint were disease-specific survival (DSS) and overall survival (OS). Further secondary endpoints were the assessment of IFN tolerability in post-surgical patients and the observation of prognostic factors related to early or late recurrence. Adherent patients were considered for a subgroup analysis focused on patients who effectively received the treatment designed to prevent HCC recurrence.

Enrolment for the trial started on June 1998. By December 2002 the predicted sample size of 150 randomized patients was completed ("pure HCV": 80 and "mixed HCV+HBV": 70). The baseline clinical, laboratory and tumor characteristics of the two arms and viral strata were comparable. After 45 months of median follow-up the three- and five- years survival rates were 69% and 52.4% respectively for the control group and 77.3% and 63.6% respectively for the IFN group (P= 0.471) . At the univariate analysis tumor multiplicity (>1 nodule) and vascular invasion were significantly related to recurrence. After adjustment of the relative weight of prognostic factors in a series of Cox models and cumulative incidence curves calculated on pattern of recurrence, a benefit of IFN was observed on late recurrence occurring in the pure-HCV patients adherent to treatment (hazard rate: 0.3; 95% Confidence interval:0.09-0.9, P=0.04).

In conclusion, although adjuvant IFN failed to show a generalized effect on prevention of HCC recurrence after curative resection, it effectively reduced late recurrence due to new tumor foci in pure-HCV patient adherent to therapy (i.e.: receiving at least 80% of IFN dose for at least 80% of time).

ELIGIBILITY:
Inclusion Criteria:

* HCV-RNA positive / HBsAg-negative patients with HCC undergoing potentially curative resection
* Curative surgery (i.e. no residual tumor intraoperative US and tumor-free margins at pathology)
* No recurrence 1 month after surgery (CT, NMR, US)
* Pre-resection treatments allowed (TACE, RFA, PEI)
* HCV-RNA positive (lower limit of detection: 100 copies/ml) regardless of blood titers or genotype

Exclusion Criteria:

* HBsAg-positivity
* Evidence of any active neoplastic site
* Previous IFN or chemotherapy or treatment of other tumors
* Severe surgical complication and/or causes of cirrhosis not related to HCV
* Patient comorbidity (Hb <12 g/dl, HIV infection, autoimmune disease, psychiatric disorder, seizure, severe cardiovascular disease, poorly controlled diabetes, BMI >35)
* Active alcohol intake (>80 g/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 1998-06; Study Completion 2005-09

PRIMARY OUTCOMES:
Recurrence Free Survival

SECONDARY OUTCOMES:
Disease Specific Survival
Overall Patient Survival

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, Principal Investigator — National Cancer Institute, Milan, Italy
Locations (1):
- National Cancer Institute, Milan, Italy

REFERENCES:
- [Derived] Mazzaferro V, Romito R, Schiavo M, Mariani L, Camerini T, Bhoori S, Capussotti L, Calise F, Pellicci R, Belli G, Tagger A, Colombo M, Bonino F, Majno P, Llovet JM; HCC Italian Task Force. Prevention of hepatocellular carcinoma recurrence with alpha-interferon after liver resection in HCV cirrhosis. Hepatology. 2006 Dec;44(6):1543-54. doi: 10.1002/hep.21415. PMID 17133492